CLINICAL TRIAL: NCT04699409
Title: The Comparison of Educational Effectiveness Between FAST and STROKE 112 in Yunlin Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202009041RIND
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Stroke, Cardiovascular
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAST (Experimental): stroke education: FAST
  Interventions: Other: stroke educational campaign: FAST
- STROKE 112 (Experimental): stroke education: STROKE 112
  Interventions: Other: stroke educational campaign: STROKE 112

INTERVENTIONS:
Other: stroke educational campaign: FAST — After randomization, study staff provided 15-minute education on the selected campaign to each individual participant using educational pictures.
  Arms: FAST
Other: stroke educational campaign: STROKE 112 — After randomization, study staff provided 15-minute education on the selected campaign to each individual participant using educational pictures.
  Arms: STROKE 112

SUMMARY:
FAST and Stroke-112 are two campaigns to reduce the emergency room arrival time of stroke patients. No study has evaluated the effectiveness of these campaigns. This study aimed to compare recalling capacity of people in these two campaigns.

DETAILED DESCRIPTION:
Cerebral vascular accidents have been one of the leading causes of death in Taiwan in recent years. In the modern medical system, treatment for hyperacute stroke including intravenous thrombolysis and intra-arterial thrombectomy. The faster patient received treatment, the better outcome he has.

Prehospital delay of acute stroke treatment has been an important issue in modern medical system. Awareness of stroke symptoms and calling for medical help immediately is the most important part of stroke health education. The most used educational campaign is FAST.

In recent years, there is another stroke educational campaign called STROKE 112. Previous study had showed it has greater acceptance, since the number is easier to remember then letter, especially in non-English speaking countries.

The investigators had conducted a hospital-based randomized study in 2019, which revealed that STROKE 112 had similar, but not superior effectiveness with FAST. However, more study is needed for community-based population.

This study will compare and explore the effectiveness of two stroke educational campaigns, FAST and STROKE 112, on community-based population by using the questionnaire, in Yunlin, Taiwan. The result will been compared and analyzed with previous study, help us modify and enhance our current stroke educational program, shorten the prehospital delay, and improve outcomes of patients with acute stroke.

The subjects will be randomized into either group: FAST or STROKE 112. Then the investigator will give a 15min eduacation. The evaluation will be arranged 5 days and 30 days after the first education, and the outcome is the recalling capacity of the stroke symptoms in the educational campaign.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20
* individuals who could speak either Mandarin or Taiwanese as their mother tongue

Exclusion Criteria:

* individuals who could not understanding the education campaign(ex. dementia, aphasia)
* individuals who were previously aware about either campaign

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The recalling capacity of the stroke symptoms mentioned in each campaign | 5 days
  Compare recalling capacity of people in these two campaigns: uneven face, weak arm, slurred speech. If the patient could recall one symptom, then he get 1 score. Total score is 3(which means the subject can recall all three symptoms)
The recalling capacity of the stroke symptoms mentioned in each campaign | 30 days
  Compare recalling capacity of people in these two campaigns: uneven face, weak arm, slurred speech. If the patient could recall one symptom, then he get 1 score. Total score is 3(which means the subject can recall all three symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: YiTe Tsai, Bachelor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD